CLINICAL TRIAL: NCT04117906
Title: Developing and Piloting an Online, Self-help Intervention for Anxiety
Brief Title: Developing and Piloting an Online, Self-help Intervention (STAGE) for Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AsukaBoyleMRP2017
Record Dates: First submitted 2019-10-04; First posted 2019-10-07 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2019-10

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Measures will be completed online without direct involvement from the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STAGE course (Experimental)
  Interventions: Behavioral: STAGE training for anxiety
- Wait-list control (No Intervention): The wait-list control group will receive access to the STAGE course after the trial is complete.

INTERVENTIONS:
Behavioral: STAGE training for anxiety — STAGE is a brief, online, self-help course designed to target anxiety through providing training in perspective broadening and self-distancing.
  Arms: STAGE course

SUMMARY:
This study pilots a novel, brief, online, self-help training course for anxiety management, aimed at adults experiencing moderate to moderately-severe anxiety.

DETAILED DESCRIPTION:
This study is a pilot randomised controlled trial (RCT) comparing a brief, online self-help, anxiety management training course ('STAGE') with a wait-list control. A battery of self-report measures will be administered online at baseline (week 0), post-intervention (week 3) and at follow-up (week 5).

ELIGIBILITY:
Inclusion Criteria:

* having a score, at baseline, on the Generalised Anxiety Disorder 7 (GAD-7) scale of between 8 and 15, inclusive;
* having regular internet access;
* being based in the UK.

Exclusion Criteria:

* significant risk issues in the last year;
* currently receiving another psychological intervention, whether it be self-help or face-to-face;
* having recently (within the last six months) completed a psychological intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline (week 0) at post-intervention (week 3) on the Generalised Anxiety Disorder 7 (GAD-7) scale. | Post-intervention (3 weeks after baseline).
  The Generalised Anxiety Disorder 7 (GAD-7) scale is a self-report measure of general anxiety, producing a total score between 0 and 21, with higher scores indicating greater levels of general anxiety.

SECONDARY OUTCOMES:
Change from baseline (week 0) at follow-up (week 5) on the Generalised Anxiety Disorder 7 (GAD-7) scale. | Follow-up (5 weeks after baseline).
  As described above
Change from baseline (week 0) at post-intervention (week 3) on the Patient Health Questionnaire 9 (PHQ-9). | Post-intervention (3 weeks after baseline).
  The Patient Health Questionnaire 9 (PHQ-9) is a self-report measure of depression, producing a total score between 0 and 27, with higher scores indicating greater levels of depression.
Change from baseline (week 0) at follow-up (week 5) on the Patient Health Questionnaire 9 (PHQ-9). | Follow-up (5 weeks after baseline).
  As described above
Change from baseline (week 0) at post-intervention (week 3) on the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). | Post-intervention (3 weeks after baseline).
  The Warwick-Edinburgh Mental Well-Being Scale (WEMWBS) is a self-report measure of mental wellbeing, producing a total score between 14 and 70, with higher scores indicating greater levels of mental wellbeing.
Change from baseline (week 0) at follow-up (week 5) on the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS). | Follow-up (5 weeks after baseline).
  As described above
Change from baseline (week 0) at post-intervention (week 3) on the Experience Questionnaire (EQ). | Post-intervention (3 weeks after baseline).
  The Experience Questionnaire (EQ) is a self-report measure of decentering, producing a total score between 20 and 100, with higher scores indicating greater levels of decentering.
Change from baseline (week 0) at follow-up (week 5) on the Experience Questionnaire (EQ). | Follow-up (5 weeks after baseline).
  As described above
Change from baseline (week 0) at post-intervention (week 3) on the Putting into Perspective subscale of the Cognitive Emotion Regulation Questionnaire (CERQ). | Post-intervention (3 weeks after baseline).
  The Putting into Perspective subscale of the Cognitive Emotion Regulation Questionnaire (CERQ) is a self-report measure of perspective taking, producing a total score between 4 and 20.
Change from baseline (week 0) at follow-up (week 5) on the Putting into Perspective subscale of the Cognitive Emotion Regulation Questionnaire (CERQ). | Follow-up (5 weeks after baseline).
  As described above

CONTACTS AND LOCATIONS:
Overall Officials: Asuka Boyle, MSc, Principal Investigator — Canterbury Christ Church University; Fergal Jones, PhD, PsychD, Study Director — Canterbury Christ Church University; Emma Travers-Hill, PhD, PsychD, Study Director — Kent and Medway NHS and Social Care Partnership Trust
Locations (1):
- Canterbury Christ Church University, Royal Tunbridge Wells, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No